CLINICAL TRIAL: NCT05158374
Title: Molecular Effects of Aspirin & Metformin on Colonic Epithelium
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn prior to gaining approvals
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: AC21120
Record Dates: First submitted 2021-11-17; First posted 2021-12-15 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Control (No Intervention): No medication, 6 weeks
- Aspirin 24 Hours (Active Comparator): 24 Hours Aspirin
  Interventions: Drug: Aspirin tablet
- Aspirin 7 Days (Active Comparator): 7 Days Aspirin
  Interventions: Drug: Aspirin tablet
- Aspirin 28 Days (Active Comparator): 28 Days Aspirin
  Interventions: Drug: Aspirin tablet
- Aspirin 6 Weeks (Active Comparator): 6 Weeks Aspirin
  Interventions: Drug: Aspirin tablet
- Metformin 24 Hours (Active Comparator): 24 Hours Metformin
  Interventions: Drug: Metformin
- Metformin 7 Days (Active Comparator): 7 Days Metformin
  Interventions: Drug: Metformin
- Metformin 28 Days (Active Comparator): 28 Days Metformin
  Interventions: Drug: Metformin
- Metformin 6 Weeks (Active Comparator): 6 Weeks Metformin
  Interventions: Drug: Metformin
- Aspirin & Metformin 24 Hours (Active Comparator): 24 Hours Aspirin & Metformin
  Interventions: Drug: Aspirin and Metformin
- Aspirin & Metformin 7 Days (Active Comparator): 7 Days Aspirin & Metformin
  Interventions: Drug: Aspirin and Metformin
- Aspirin & Metformin 28 Days (Active Comparator): 28 Days Aspirin & Metformin
  Interventions: Drug: Aspirin and Metformin
- Aspirin & Metformin 6 Weeks (Active Comparator): 6 Weeks Aspirin & Metformin
  Interventions: Drug: Aspirin and Metformin

INTERVENTIONS:
Drug: Aspirin tablet — 75mg Aspirin once per day
  Other Names: acetylsalicylic acid
  Arms: Aspirin 24 Hours; Aspirin 28 Days; Aspirin 6 Weeks; Aspirin 7 Days
Drug: Metformin — 500mg Metformin once per day
  Other Names: Glucophage
  Arms: Metformin 24 Hours; Metformin 28 Days; Metformin 6 Weeks; Metformin 7 Days
Drug: Aspirin and Metformin — 75mg Aspirin and 500mg Metformin once per day
  Other Names: acetylsalicylic acid and Glucophage
  Arms: Aspirin & Metformin 24 Hours; Aspirin & Metformin 28 Days; Aspirin & Metformin 6 Weeks; Aspirin & Metformin 7 Days

SUMMARY:
Bowel cancer, a significant problem in the United Kingdom (UK) with ~ 41,000 diagnoses and ~ 16,000 deaths annually, has a large preventable component (~54%). It is, in part, due to energy imbalance within bowel cells as suggested by associated risk factors: high-fat diet, obesity, physical inactivity and type 2 diabetes mellitus. Drugs that decrease bowel cancer risk, like aspirin and metformin, may prevent the disease by mimicking the molecular effects of dietary restriction and exercise.

Energy imbalance, through obesity, expands stem cells which may increase bowel cancer. We have shown that aspirin activates an energy molecule, which increases when we exercise, and blocks signalling associated with obesity in bowel cancer. Indeed aspirin in combination with metformin (commonly used in diabetes) has a greater effect on this pathway than either drug alone.

To predict which patients may benefit from aspirin and metformin, we need to discover if these drugs may mimic healthy lifestyle changes at a cellular level and which cells are being targeted.

This project investigates how aspirin and metformin influence energy molecules in bowel cells to mimic beneficial effects of exercise or dietary restriction. Participants, recruited from Western General Hospital (Edinburgh) colorectal clinics, will have bowel lining and blood samples take initially and then depending on their assigned cohort, after; 24 hours, 7 days, 28 days or a 6-week course of aspirin, metformin or both tablets. Samples will be analysed for energy genes (main outcome). Secondary outcomes will measure effects on quantitative faecal immunochemical tests (qFIT), used to detect blood in the stool, and on gut bacteria.

This critical research will inform how aspirin and metformin can be used in specific populations to decrease bowel cancer risk and to develop new drugs to target abnormal energy pathways.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is eminently preventable, and yet it is the 2nd most common cause of cancer death in the UK. Both population growth and ageing will influence CRC incidence. There is a significant environmental aetiological component, with around 54% being preventable. Modifiable risk factors include obesity, metabolic syndrome, type 2 diabetes mellitus (T2DM), and physical inactivity.Recent data suggests that the rising CRC incidence in young populations is associated with the increase in obesity and T2DM. Hence, there is substantial rationale for developing approaches that define and modify CRC obesity-related risk. Cancer cells have long been observed to reprogramme metabolism to generate substrates for growth. There are multiple molecular mechanisms linking obesity and CRC. Obesity is the commonest cause of insulin resistance and T2DM. Obesity-mediated insulin resistance and inflammation may drive CRC. Obesity increases early CRC precursor lesions of aberrant crypt foci. Bariatric surgery reduces adenomas and decreases CRC risk biomarkers such as proliferation and inflammation markers. High-fat diet (HFD) animal models of obesity and carcinogen-induced CRC show intestinal stem cell expansion. Dietary fatty acids themselves may drive stem cell expansion. Highlighting further complexity, intestinal epithelial insulin receptor deletion attenuates the HFD-induced increase in cholesterol and stem cell messenger ribonucleic acids (mRNAs).

Calorie restriction, associated with longevity and reduced cancer incidence, may be mediated through downregulation of nutrient-sensing pathways. Agents that clearly decrease CRC incidence, such as aspirin and metformin (may act as calorie restriction mimetics by influencing nutrient-sensing. The host lab have shown that low-dose aspirin reduces CRC incidence in the Scottish population and that high-energy snacks are associated with CRC risk -strengthening the link between energy, diet and cancer. They also demonstrated that aspirin modulates key nutrient-sensing pathways; aspirin activates AMP-activated protein kinase (AMPK) and inhibits mammalian target of rapamycin (mTOR) signalling in CRC cells, mouse intestine and patients. Furthermore, there was a synergistic effect with aspirin and metformin with respect to AMPK activation and mTOR inhibition in CRC cells. The protective effect of aspirin may be greater in higher body-mass index (BMI) patients. Mendelian randomisation studies strengthen causal links between obesity, hyperlipidaemia, pro-inflammatory fatty acids and CRC risk.

This study aims to elucidate the underlying molecular mechanisms of aspirin and metformin with respect to their cancer preventing properties in the colon, thereby identifying potential critical "druggable" targets. The ultimate aim is to predict which patients may benefit from these drugs to prevent CRC.

ELIGIBILITY:
Inclusion Criteria:

All participants who are capable of giving informed consent. All participants aged 16 years or over. All participants must have no known contraindications to rectal biopsy procedures.

All participants must be resident in the United Kingdom. All participants must have no known contraindications to aspirin and metformin.

Exclusion Criteria:

Unable to give informed consent. Under the age of 16 years. Individuals who are taking anti-coagulation medication. Individuals with platelet disease or other bleeding issues. Individuals with a history of a significant rectal bleed. History of diabetes mellitus or impaired glucose tolerance. Any contraindication to either aspirin or metformin. Female subjects of child bearing age who are not taking effective contraception during the period of the trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 24 hours Aspirin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 7 days Aspirin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 28 days Aspirin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 6 weeks Aspirin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 24 hours Metformin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 7 days Metformin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 28 days Metformin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 6 weeks Metformin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 24 hours combined Aspirin and Metformin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 7 days combined Aspirin and Metformin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 28 days combined Aspirin and Metformin medication
  Effect on genetic expression
Relative genetic expression change of genes relating to energy, metabolism and stem cell signalling in the large bowel | Baseline and immediately after 6 weeks combined Aspirin and Metformin medication
  Effect on genetic expression

SECONDARY OUTCOMES:
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 24 hours Aspirin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 7 days Aspirin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 28 days Aspirin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 6 weeks Aspirin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 24 hours Metformin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 7 days Metformin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 28 days Metformin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 6 weeks Metformin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 24 hours Aspirin and Metformin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 7 days Aspirin and Metformin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 28 days Aspirin and Metformin medication
  Effect of qFIT value
Change in value of qFIT result with aspirin, metformin or combination | Baseline and immediately after 6 weeks Aspirin and Metformin medication
  Effect of qFIT value
Change in the proportions of bacterium in the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 24 hours Aspirin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 7 days Aspirin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 28 days Aspirin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 6 weeks Aspirin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 24 hours Metformin medication
  Effect on microbiome
Change in the proportions of bacterium colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 7 days Metformin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 28 days Metformin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 6 weeks Metformin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 24 hours Aspirin and Metformin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 7 days Aspirin and Metformin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 28 days Aspirin and Metformin medication
  Effect on microbiome
Change in the proportions of bacterium the colorectal microbiome after aspirin and/or metformin medication | Baseline and immediately after 6 weeks Aspirin and Metformin medication
  Effect on microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Farhat VN Din, FRCSed, Principal Investigator — University of Edinburgh

IPD SHARING:
Plan to Share IPD: No